CLINICAL TRIAL: NCT04418362
Title: Axon - Brain Train for Pain - A Home-based Neurofeedback Intervention to Treat the Primary and Secondary Symptoms of Chronic Pain
Brief Title: Axon - Brain Train for Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Exsurgo Rehab Limited (Industry)
Collaborators: East Midlands Spine Ltd (Unknown); PhysioFunction Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ED1001033
Record Dates: First submitted 2020-05-29; First posted 2020-06-05 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2020-07

CONDITIONS: Chronic Pain; Depression, Anxiety; Sleep; Quality of Life
MeSH Terms: conditions — Chronic Pain; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurofeedback training (Experimental): Neurofeedback training: self-administered at home 4-6 times per week for 8 weeks. Each session consists of 6 blocks of 5 minute training with a one minute rest period between each block.
  Interventions: Other: Neurofeedback training

INTERVENTIONS:
Other: Neurofeedback training — A home-based self-administered neurofeedback intervention taking place 4-6 times per week for 8 weeks.

SUMMARY:
A mixed methods proof of concept study to ascertain the effectiveness of a home-based self-administered neurofeedback intervention to treat the primary and secondary symptoms of chronic pain.

DETAILED DESCRIPTION:
In order to address the growing problem of chronic pain management in the UK, a proof of concept/feasibility open label study has been devised to test a home-based self-administered non-pharmacological treatment utilising neurofeedback training with a headset and tablet-based software application.

This study will include individuals suffering from various types of chronic pain, measuring changes in pain intensity alongside associated symptoms (depression, anxiety, sleep, and quality of life) by utilising a purpose-built software application and headset that is easy to use and structurally robust.

Twenty participants will take part in pre-intervention quantitative assessments measuring the primary and secondary symptoms of chronic pain. This will be followed by one-to-one remote training where they will be provided with detailed instructions on how to self-administer the neurofeedback training in the comfort of their own homes. They will then take part in 4-6 training sessions per week over an 8-week period.

Post- intervention quantitative assessments will be conducted alongside a qualitative analysis of the experience of doing neurofeedback training for chronic pain. Participant feedback on how the protocol, equipment and research could be improved will also be recorded to inform further research.

Participants will also take part in online follow-up assessments at 1, 3, and 6 months after the intervention. Any adjustments to pain medication will also be recorded over this period. It is anticipated this study will provide initial evidence of the safety, efficacy, reliability and validity of a low-cost non-pharmacological solution to the physical, psychological and social difficulties experienced by individuals with chronic pain, with a view to a larger subsequent multisite trial.

ELIGIBILITY:
Inclusion Criteria:

* Head circumference range (560 - 595 mm)
* Patients suffering from chronic pain (mean VNS >4) for at least 6 months.
* Chronic pain from any neurological or musculoskeletal cause, of which examples could be, post herpetic (or post-shingles) neuralgia, complex regional pain syndrome (CRPS), lower back pain, neck pain, major joint pain, spinal cord injury, phantom limb pain, brachial plexus injury related pain, traumatic peripheral nerve injury pain and post-cancer treatment pain
* Stable medication and treatment over the intervention period
* Participant or caregiver with minimum computer literacy able to effectively operate equipment after training, and the ability to position and remove headset effectively for training sessions

Exclusion Criteria:

* Patients who do not meet inclusion criteria (above)
* Failing pre-screening suitability criteria for neurofeedback due to a neurological disorder, psychiatric disorder, epilepsy, regular use of benzodiazepines, previous neurofeedback training, serious head injury and other medication that has contraindications for neurofeedback training
* Dreadlocks, braids, beads, or any other hairstyle or hair covering that cannot be removed for training
* Known or suspected pregnancy
* Diagnosis of (or currently undergoing treatment for) cancer, systemic infection, severe cardiovascular/respiratory comorbidity
* Implanted electronic neuromodulation device
* Implanted pacemaker or loop recorder
* Any change in medication or treatment planned during the intervention period
* Inability to use the equipment due to severity of pain

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-07-28 (Actual)

PRIMARY OUTCOMES:
Change in pain intensity as measured by the VNS (Visual Numerical Scale) | Pre-intervention, before and after each training session over 8 week period, and 1, 3 and 6 months after final training session
  Ordinal measurement of individual's pain intensity

SECONDARY OUTCOMES:
Change in mood as measured by Hospital Anxiety and Depression Scale (HADS) | Pre-intervention, after the final training session (8 weeks), and 1, 3 and 6 months after final session
  Rating scale (self-administered)
Change in quality of sleep as measured by the Pittsburgh Sleep Quality Index (PSQI) | Pre-intervention, after the final training session (8 weeks), and 1, 3 and 6 months after final session
  A self-report questionnaire assessing sleep quality
Change in quality of life components as measured by the EQ-5D-5L | Pre-intervention, after the final training session (8 weeks), and 1, 3 and 6 months after final session
  A self-assessed, health related, quality of life questionnaire.
Changes in EEG activity | Baseline (eyes open and eyes closed) pre-intervention, and before and after each training session over 8 weeks
  Changes in relative Alpha, Theta and Beta ratio, as measured by EEG
Experience of chronic pain and neurofeedback training | Post-intervention - after final training session (8 weeks)
  Qualitative interviews of the lived experience of taking part in neurofeedback training for chronic pain

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Birch, Principal Investigator — East Midlands Spine Ltd
Locations (1):
- East Midlands Spine Ltd, Northampton, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Birch N, Graham J, Ozolins C, Kumarasinghe K, Almesfer F. Home-Based EEG Neurofeedback Intervention for the Management of Chronic Pain. Front Pain Res (Lausanne). 2022 May 27;3:855493. doi: 10.3389/fpain.2022.855493. eCollection 2022. PMID 35712448